CLINICAL TRIAL: NCT04292002
Title: Test@Work: Evaluation of Attitudes and Uptake Within Employee Health Checks in the Construction Industry
Brief Title: Test@Work Study: Evaluation of Attitudes and Uptake Within Employee Health Checks in the Construction Industry
Acronym: Test@Work
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Holly Blake, Associate Professor of Behavioural Science, University of Nottingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IN-UK-276-5347 HIV DVE
Record Dates: First submitted 2019-12-06; First posted 2020-03-02 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: HIV
Keywords: workplace; health promotion; health screening; employees; health behaviour

STUDY DESIGN:
Intervention Model Description: The investigators are looking at uptake and reach of general health checks offered to up to 650 employees in the construction industry.
Masking Description: Not relevant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health Checks (Experimental): Workplace health checks - in this intervention employees can select from a range of optional health checks/tests and receive tailored health advice and a health resource pack.
  Interventions: Behavioral: Test@Work

INTERVENTIONS:
Behavioral: Test@Work — Offer of a general health check including opt-in sexual health consultation and HIV testing, weight/height, Body Mass Index (BMI), blood pressure, mental health screen. Provision of tailored health advice and a resource pack with information and signposting.

SUMMARY:
This project is called Test@Work. In this project the investigators will offer general health checks and tailored health advice to up to 650 employees in the construction industry at sites across the East Midlands. The investigators will assess reach and uptake, and evaluate the views and perceptions of employees, managers and the delivery team. Health checks will include Body Mass Index (BMI; weight/height), waist-to-hip ratio, blood pressure, mental health screen, sexual health consultation and an opt-in rapid screening test for human immunodeficiency virus (HIV). Employees will be provided with a resource pack with information and signposting around physical activity, diabetes risk, diet, and musculoskeletal health. A digital resource providing information and signposting about workplace health screening and HIV testing will be developed and provided to managers at the participating worksites 2 weeks before their health check event.

Employees will be offered an additional text messaging service involving receipt of a series of messages with advice around HIV and testing alongside general health information. Employees will complete post-health check exit questionnaires and an exit interview. Managers will complete a post-event evaluation questionnaire and post-event interview. Mixed-methods evaluation will include assessment of reach, uptake, and intervention implementation processes.

DETAILED DESCRIPTION:
The investigators will collect evaluation data with employees and company representatives.

Employees: will complete exit-questionnaires and be invited to a brief exit interview.

The investigators will collect by anonymous questionnaire: age, gender, country of birth, ethnicity, postcode, sexual orientation, employment status (FT/PT, permanent, agency, contract worker), reasons for attending, health perceptions, prior HIV testing history, influence of work on health, perceptions of employers provision for health and wellbeing, perceptions towards HIV testing in the workplace, range of tests undertaken, views about the workplace health check and future health intentions. Personal identifiers will not be collected and questionnaire data will not be provided to employers. Those employees who agree to be interviewed after the health check will be invited to a brief independent confidential interview with the project researcher.

Company representatives: will complete brief post-event questionnaire and be invited to post-event interview

The investigators will ask about the organisational/employee profile, their perceptions of company provision for health and wellbeing, perceptions towards the usefulness of the implementation toolkit and towards HIV testing in the workplace, method of delivery and their confidence to support employees who disclose a positive test outcome, views about the workplace health check and future implementation intentions.

ELIGIBILITY:
Inclusion Criteria:

* employee of a company in construction or related industries
* provides informed consent

Exclusion Criteria:

* does not speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 456 (Actual)
Dates: Start 2019-08-17 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Health check uptake | Rolling intervention delivery and data collection over 15 months
  Percentage of employees choosing to take a workplace health check from total employee population across all sites

SECONDARY OUTCOMES:
reasons for attending | immediately post-event
  Qualitative data collected on reasons for opting in to health check
perceptions of employer's provision for health and wellbeing | immediately post-event
  Qualitative data collected on perceptions towards employer
perceptions towards HIV testing in the workplace | immediately post-event
  Qualitative data collected on employee views towards HIV testing at work
range of tests undertaken | during the health check, and qualitative data immediately post-event
  which of the optional checks/tests were taken by the employee
Employee demographic profile | At recruitment
  Age, Gender, country of birth, ethnicity, postcode, sexual orientation, employment status (full-time or part-time, permanent, agency, contract worker)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nottingham, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The investigators are not collecting individual health outcomes as part of this study. The primary aim is to assess uptake and reach of this workplace health checks initiative. Anonymised qualitative data can be available on reasonable request.

REFERENCES:
- [Background] Blake H, Somerset S, Evans C. Development and Fidelity Testing of the Test@Work Digital Toolkit for Employers on Workplace Health Checks and Opt-In HIV Testing. Int J Environ Res Public Health. 2020 Jan 6;17(1):379. doi: 10.3390/ijerph17010379. PMID 31935985
- [Result] Blake H, Somerset S, Whittingham K, Middleton M, Yildirim M, Evans C. WHIRL Study: Workplace Health Interprofessional Learning in the Construction Industry. Int J Environ Res Public Health. 2020 Sep 18;17(18):6815. doi: 10.3390/ijerph17186815. PMID 32961985
- [Result] Middleton M, Somerset S, Evans C, Blake H. Test@Work Texts: Mobile Phone Messaging to Increase Awareness of HIV and HIV Testing in UK Construction Employees during the COVID-19 Pandemic. Int J Environ Res Public Health. 2020 Oct 26;17(21):7819. doi: 10.3390/ijerph17217819. PMID 33114546
- [Result] Somerset S, Evans C, Blake H. Accessing Voluntary HIV Testing in the Construction Industry: A Qualitative Analysis of Employee Interviews from the Test@Work Study. Int J Environ Res Public Health. 2021 Apr 15;18(8):4184. doi: 10.3390/ijerph18084184. PMID 33920943
- [Derived] Jones W, Somerset S, Evans C, Whittingham K, Middleton M, Blake H. Test@work: evaluation of workplace HIV testing for construction workers using the RE-AIM framework. BMC Public Health. 2021 Sep 24;21(1):1737. doi: 10.1186/s12889-021-11739-z. PMID 34560853
- See also: news item — https://www.nottingham.ac.uk/healthsciences/news/workplace-health-innovation-construction-industry.aspx
- See also: news item — http://www.theconstructionindex.co.uk/news/view/breaking-the-hiv-taboo